CLINICAL TRIAL: NCT00472745
Title: Nutritional Regulation of Bone - Pilot Study
Brief Title: The Effect of Weight Loss on Bone in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Sue A. Shapses, Ph.D., RD, Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG0084; 5R01AG012161 (NIH)
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2022-01

CONDITIONS: Weight Loss; BMD
Keywords: bone mass; calcium absorption; bone quality; fracture risk; arthritis; osteoporosis
MeSH Terms: conditions — Weight Loss; Arthritis; Osteoporosis | interventions — Body Weight Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WL (Experimental): weight loss (WL) with nutrition/behavior modification counseling
  Interventions: Behavioral: Weight Loss
- WM (Active Comparator): Weight Maintenance (WM)
  Interventions: Behavioral: Weight Maintenance

INTERVENTIONS:
Behavioral: Weight Loss — Weight loss participants will consume a reduced calorie diet based on their individual caloric needs to lose 1.5-2 lbs/week, and will attend regular counseling sessions (for about 45 minutes each) with a dietitian for 6 months
  Arms: WL
Behavioral: Weight Maintenance — Diet for weight maintenance for 6 months
  Arms: WM

SUMMARY:
The purpose of this study is to determine the effect of weight loss on bone health in men.

DETAILED DESCRIPTION:
This pilot study of the effect of weight loss on bone health in men is being undertaken in conjunction with studies of the effect of weight loss on bone health in women for comparison purposes. See NCT00473031, NCT00472680, and NCT00472654. This information is important for determining optimal nutrient requirements during weight loss.

Participants will be recruited for both weight loss and weight maintenance. All participants will be asked to take a daily vitamin/mineral supplement and, depending on their usual food intake, they may be asked to take a calcium tablet to meet the recommended intake throughout the study period. Weight loss participants will attend regular counseling sessions (about 45 minutes each) with a dietitian for approximately 6 months; they will be asked to attend 6 sessions but will be given the opportunity to attend 13 sessions. Body composition will be measured by a dual-energy x-ray absorptiometry (DXA) machine, ultrasound, and peripheral quantitative computer tomography (pQCT) before and after 6 months of weight loss. Bone, mineral, protein and lipid markers, and hormones that influence bones will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Obese or overweight
* Must live in the geographic vicinity of Rutgers University

Exclusion Criteria:

* Currently on any medication known to influence calcium or bone metabolism, including HRT, or with evidence of diseases known to influence calcium metabolism (i.e. metabolic bone disease, hyperparathyroidism, untreated thyroid disease, significant immune, hepatic, or renal disease, significant cardiac disease [i.e., heart attack or stroke in the past 6 months., abnormal EKG], active malignancy or cancer therapy within the past year)
* History of kidney stones
* Weight gain or weight loss (5% of body wt) within 3 months prior to recruitment
* Participation in other investigational studies during the 12-month study period
* Usually have a very high or low intake of calcium (more than 1500 or less than 500 mg per day)

Ages: 50 Years to 72 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Changes in bone density and quality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sue Shapses, PhD, RD, Principal Investigator — Rutgers University, Nutritional Sciences
Locations (1):
- Rutgers University, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Shapses SA, Riedt CS. Bone, body weight, and weight reduction: what are the concerns? J Nutr. 2006 Jun;136(6):1453-6. doi: 10.1093/jn/136.6.1453. PMID 16702302
- [Background] Riedt CS, Cifuentes M, Stahl T, Chowdhury HA, Schlussel Y, Shapses SA. Overweight postmenopausal women lose bone with moderate weight reduction and 1 g/day calcium intake. J Bone Miner Res. 2005 Mar;20(3):455-63. doi: 10.1359/JBMR.041132. Epub 2004 Nov 29. PMID 15746990
- [Background] Cifuentes M, Riedt CS, Brolin RE, Field MP, Sherrell RM, Shapses SA. Weight loss and calcium intake influence calcium absorption in overweight postmenopausal women. Am J Clin Nutr. 2004 Jul;80(1):123-30. doi: 10.1093/ajcn/80.1.123. PMID 15213038
- [Background] Goode LR, Brolin RE, Chowdhury HA, Shapses SA. Bone and gastric bypass surgery: effects of dietary calcium and vitamin D. Obes Res. 2004 Jan;12(1):40-7. doi: 10.1038/oby.2004.7. PMID 14742841
- [Background] Pop LC, Sukumar D, Tomaino K, Schlussel Y, Schneider SH, Gordon CL, Wang X, Shapses SA. Moderate weight loss in obese and overweight men preserves bone quality. Am J Clin Nutr. 2015 Mar;101(3):659-67. doi: 10.3945/ajcn.114.088534. Epub 2015 Jan 7. PMID 25733651
- [Derived] Ogilvie AR, Schlussel Y, Sukumar D, Meng L, Shapses SA. Higher protein intake during caloric restriction improves diet quality and attenuates loss of lean body mass. Obesity (Silver Spring). 2022 Jul;30(7):1411-1419. doi: 10.1002/oby.23428. Epub 2022 May 11. PMID 35538903